CLINICAL TRIAL: NCT06196619
Title: The Relationship of Shear Wave Elastography Findings With Pain Threshold and Quality of Life in Patients With Lipedema
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: gulcanozturkchatip
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-11

CONDITIONS: Pain; Lipedema
Keywords: Shear Wave Elastography; Pain; Lipedema
MeSH Terms: conditions — Pain; Lipedema | interventions — Visual Analog Scale

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stage 1 lipedema patients: It is the stage where normal skin surface, enlarged subcutaneous fat tissue, and many small nodules are present upon palpation.
  Interventions: Diagnostic Test: SWE:B-mode ultrasound and subcutaneous elastic modulus with shear wave elastography at three level
- Stage 2 lipedema patients: It is the stage with rough skin surface, large nodules of palpable subcutaneous fat tissue
  Interventions: Diagnostic Test: SWE:B-mode ultrasound and subcutaneous elastic modulus with shear wave elastography at three level
- Stage 3 lipedema patients: It is the stage in which lobular deformation of the skin surface occurs with enlarged fatty tissue.
  Interventions: Diagnostic Test: SWE:B-mode ultrasound and subcutaneous elastic modulus with shear wave elastography at three level

INTERVENTIONS:
Diagnostic Test: SWE:B-mode ultrasound and subcutaneous elastic modulus with shear wave elastography at three level — Visual analog scale(VAS):This scale measure in which individuals rate their pain from 0 to 10, with 0 indicating no pain at all and 10 representing the worst pain;pain threshold through algometric measurement; quality of life using the EQ-5D general quality of life scale.
  Other Names: visual analog scale(VAS); pain threshold through algometric measurement; EQ-5D general quality of life scale.

SUMMARY:
The aim of this study is to evaluate the relationship between disease severity and subcutaneous tissue shearwave elastography findings with pain threshold and quality of life in patients diagnosed with lipedema.

DETAILED DESCRIPTION:
Patients diagnosed with lipedema were divided into 3 stages according to disease severity. Pain level was evaluated with visual analogue scale, pain threshold with algometric measurement, and quality of life with EQ-5D general quality of life scale. All patients underwent measurements using B-mode ultrasound and subcutaneous elastic modulus with shear wave elastography (SWE) imaging of lower limbs at three anatomical levels.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with lipedema

Exclusion Criteria:

* under 18 years of age,
* Patients with edema of cardiac or nephrogenic origin, diabetes mellitus, thyroid dysfunction, patients with lymphedema or chronic venous insufficiency, oncology patients,
* individuals with polyneuropathy, radiculopathy, or advanced degenerative diseases affecting the extremities within the last 6 months, based on clinical findings and medical history.
* patients using antiepileptics and antidepressants,
* individuals unable to cognitively tolerate participation in the study were also excluded.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study consist of female patients aged 18-70, diagnosed with lipedema
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Subcutaneous elastic modulus with shear wave elastography (SWE) imaging of lower limbs | 1 day
  Measurements using B-mode ultrasound and subcutaneous elastic modulus with shear wave elastography (SWE) imaging of lower limbs at three anatomical levels.
Visual analog scale(VAS) | 1 day
  Pain levels were assessed using the visual analog scale(VAS)
Algometric measurement | 1 day
  Pain threshold through algometric measurement
EQ-5D general quality of life scale. | 1 day
  quality of life using the EQ-5D general quality of life scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulcan Ozturk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clarke C, Kirby JN, Smidt T, Best T. Stages of lipoedema: experiences of physical and mental health and health care. Qual Life Res. 2023 Jan;32(1):127-137. doi: 10.1007/s11136-022-03216-w. Epub 2022 Aug 16. PMID 35972618
- [Background] Ishaq M, Bandara N, Morgan S, Nowell C, Mehdi AM, Lyu R, McCarthy D, Anderson D, Creek DJ, Achen MG, Shayan R, Karnezis T. Key signaling networks are dysregulated in patients with the adipose tissue disorder, lipedema. Int J Obes (Lond). 2022 Mar;46(3):502-514. doi: 10.1038/s41366-021-01002-1. Epub 2021 Nov 11. PMID 34764426
- [Background] Buso G, Depairon M, Tomson D, Raffoul W, Vettor R, Mazzolai L. Lipedema: A Call to Action! Obesity (Silver Spring). 2019 Oct;27(10):1567-1576. doi: 10.1002/oby.22597. PMID 31544340